CLINICAL TRIAL: NCT06305702
Title: Multicenter Real-world Clinical Study of Inetetamab-based Therapy in HER2-positive Metastatic Breast Cancer
Brief Title: Real-world Study of Inetetamab in HER2-positive Metastatic Breast Cancer
Status: Completed | Type: Observational
Sponsor: Liaoning Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Other Study IDs: LZRXN-001
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-02

CONDITIONS: HER2-positive Metastatic Breast Cancer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: inetetamab — 8mg/kg iv day 1 followed by 6mg/kg iv day 1, cycled every 21 days

SUMMARY:
A multicenter real-world study was conducted to gather clinicopathological data from patients with HER2-positive metastatic breast cancer who were treated with inetetamab between 2022 and 2023. The study aimed to estimate the progression-free survival (PFS), objective response rate (ORR), disease control rate (DCR), and adverse events (AEs) associated with inetetamab therapy.

ELIGIBILITY:
Inclusion Criteria:

1. An age of at least 18 years or older
2. Pathologically diagnosed with HER2-positive recurrent or metastatic breast cancer
3. Having at least one measurable lesion as defined
4. Receiving inetetamab-based therapy in the recurrent or metastatic stage
5. Having traceable medical history records

Exclusion Criteria:

1. Pregnant or lactating women
2. Patients with other conditions deemed unsuitable for participating in this study by the researcher

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HER2 Positive Advanced Breast Cancer patients who have received Inetetamab treatment in the metastatic setting.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival(PFS) | 12 months

SECONDARY OUTCOMES:
objective response rate (ORR) | 12 months
Adverse events (AEs) | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Liaoning Cancer Hospital &Institue, Shenyang, China

IPD SHARING:
Plan to Share IPD: Undecided
Our plan is to disseminate the findings of this trial via peer-reviewed articles.